CLINICAL TRIAL: NCT04059770
Title: Open Label Phase-II Randomized Trial of Three Liposomal Amphotericin B Regimens as Induction Therapy for Disseminated Histoplasmosis in AIDS Patients
Brief Title: Randomized Trial of Liposomal Amphotericin B for Histoplasmosis in AIDS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alessandro Pasqualotto (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); Hospital Nossa Senhora da Conceicao (Other); Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Sponsor-Investigator, Alessandro Pasqualotto, Principal Investigator, Federal University of Health Science of Porto Alegre
Organization: Federal University of Health Science of Porto Alegre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Three L-AmB Regimens in Histo
Record Dates: First submitted 2019-04-01; First posted 2019-08-16 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Histoplasmosis; AIDS
Keywords: Histoplasmosis; AIDS; Liposomal amphotericin B; High dose therapy
MeSH Terms: conditions — Histoplasmosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- single dose of L-AmB (Experimental): single IV dose of 10 mg/kg of L-AmB on day 1;
  Interventions: Drug: single dose of L-AmB
- 2 doses of L-AmB (Experimental): IV dose of 10 mg/kg of L-AmB on day 1, followed by 5 mg/kg of L-AmB on day 3;
  Interventions: Drug: 2 doses of L-AmB
- 2 weeks of L-AmB (Active Comparator): IV dose of 3 mg/kg of L-AmB for 2 weeks.
  Interventions: Drug: 2 weeks of L-AmB

INTERVENTIONS:
Drug: single dose of L-AmB — (i) single IV dose of 10 mg/kg of L-AmB on day 1;
  Other Names: Intervention 1
  Arms: single dose of L-AmB
Drug: 2 doses of L-AmB — (ii) IV dose of 10 mg/kg of L-AmB on day 1, followed by 5 mg/kg of L-AmB on day 3;
  Other Names: Intervention 2
  Arms: 2 doses of L-AmB
Drug: 2 weeks of L-AmB — (iii) IV dose of 3 mg/kg of L-AmB for 2 weeks.
  Other Names: Intervention 3
  Arms: 2 weeks of L-AmB

SUMMARY:
Disseminated histoplasmosis (DH) is one of the major AIDS-defining infections responsible for high mortality rates in HIV-infected patients. Liposomal amphotericin B (L-AmB) is considered the therapy of choice for AIDS-associated histoplasmosis.However, many patients in Latin America are still treated with high doses of deoxycholate amphotericin B (d-AmB) for long periods. These regimens are associated with toxicity and thus reduced efficacy. Therefore, a better treatment strategy is necessary to improve the activity of this amphotericin B treatment. Treatment with a high dose of L-AmB for short periods (rather than standard doses for longer periods) is a promising approach considering that the antifungal effect of amphotericin B depends on peak concentrations. This randomized open-label Phase II study aims to determinate and to compare the activity and safety of three L-AmB regimens, as induction therapy for DH in AIDS patients.

DETAILED DESCRIPTION:
This is a prospective randomized non-comparative multicenter open label trial of induction therapy with LAmB for DH in AIDS patients, followed by oral therapy with itraconazole.

The sample size planned is 99 patients of both sexes, older than 18 years (33 patients per study arm), infected with HIV and with confirmed diagnosis for DH. This sample size considers 10% of dropout.

The study will be conducted in accordance with the Helsinki Declaration, as well as the Standards national and international Guidelines for Good Clinical Practices.

Eight research centres in Brazil will competitively recruit patients: Santa Casa de Misericórdia de Porto Alegre (Porto Alegre; Dr Alessandro C. Pasqualotto), Hospital de Clínicas de Porto Alegre (Porto Alegre; Dr Diego R. Falci), Hospital Nossa Senhora da Conceição (Porto Alegre; Dr Marineide Melo), Hospital de Doenças Tropicais (Goiânia; Dr Cassia S. de Miranda Godoy), Hospital São José de Doenças Infecciosas (Fortaleza; Dr Terezinha M. J. Silva Leitão), and Hospital Giselda Trigueiro (Natal, Dr Monica B. Bay), Hospital Universitário Osvaldo Cruz (Recife, Dr. Filipe Prohaska Batista) e Instituto de Infectologia Emília Ribas (São Paulo, Dr. José Ernesto Vidal Bermudez).

AIDS patients with DH will be randomized to one of three study arms:

(i) single IV dose of 10 mg/kg of L-AmB; (ii) single IV dose of 10 mg/kg of L-AmB on day 1, followed by 5 mg/kg of L-AmB on day 3; (iii) IV dose of 3 mg/kg of L-AmB for 2 weeks.

Induction therapy will be followed in all patients by oral therapy with itraconazole capsules at 400 mg/daily for a year, azole drug which is already therapy of choice for consolidation of histoplasmosis, according to national and international Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years) HIV-infected hospitalized patients diagnosed with HD by the means of (i) urine Histoplasma positive antigen (IMMY® monoclonal antibody test); (ii) confirmation by classical mycological methods (microscopy, culture or histopathology); or (iii) Histoplasma positive qualitative polymerase chain reaction (PCR) in bronchoalveolar lavage samples, bone marrow aspirates or tissue samples.
* Patients will be included despite of the use of antiretroviral therapy (ART).
* Understanding and signed the Informed Consent Form.

Exclusion Criteria:

* Patients with previous diagnosis of histoplasmosis.
* Pregnant or lactating women.
* Patients with renal insufficiency (serum creatinine and urea > 1.5x the upper limit of normal).
* Abnormal aminotransferases (up to > 3x the upper limit of normal) and patients with a severe prior reaction to polyene antifungal.
* Patients who have received more than one dose of a polyene antifungal in the last 48 hours.
* Patients who refuse to participate in the study.
* Patients diagnosed with histoplasmosis that affect the central nervous system.
* Patients who, at the trial of the attending physician, are expected to die within 48 hours.
* Patients diagnosed with tuberculosis.
* Patients with any disease or condition that, in the opinion of the investigator, may interfere with the assessments or participation in the study.
* Patients receiving drugs that cause significant (relative or absolute) drug interaction with Itraconazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daiane Dalla Lana, PhD, Study Chair — Federal University of Health Science of Porto Alegre
Locations (1):
- Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Dose of L-AmB: single IV dose of 10 mg/kg of L-AmB on day 1;
  n=40
- 2 Doses of L-AmB: IV dose of 10 mg/kg of L-AmB on day 1, followed by 5 mg/kg of L-AmB on day 3;
  n=39
- 2 Weeks of L-AmB: IV dose of 3 mg/kg of L-AmB for 2 weeks.
  n=39
Period: Overall Study
Arm/Group | Single Dose of L-AmB | 2 Doses of L-AmB | 2 Weeks of L-AmB
Started | 40 | 39 | 39
Completed | 40 | 39 | 39
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10573726/pdf/ciad313.pdf
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose of L-AmB | 2 Doses of L-AmB | 2 Weeks of L-AmB | Total
Number analyzed (Participants) | 40 | 39 | 39 | 118
Age, Continuous [Median (Full Range); unit: years] | 40 [18 to 74] | 39 [18 to 74] | 39 [18 to 74] | 39 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 5 | 21
  Male | 35 | 28 | 34 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 40 | 39 | 39 | 118
Region of Enrollment [Number; unit: participants]
  Brazil | 40 | 39 | 39 | 118

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Maximum daily temperature lower than 37.8 °C
Time Frame: day 14
Population: Clinical response on day 14 was 84.0% for the single-dose L-AmB arm-(32/38-1 patient was excluded due to concomitant tuberculosis, and another was lost to follow-up), 69.0% (25/36) for the 2-dose L-AmB arm, with 3 patients being excluded from efficacy analysis (1 individual with central nervous system histoplasmosis, 1 patient with concomitant tuberculosis, and another patient lost to follow-up); in the control group, response rate was 74.0% (28/38), with 1 patient being lost to follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Single Dose of L-AmB: single IV dose of 10 mg/kg of L-AmB on day 1;
  https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10573726/pdf/ciad313.pdf
- 2 Doses of L-AmB: IV dose of 10 mg/kg of L-AmB on day 1, followed by 5 mg/kg of L-AmB on day 3;
  https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10573726/pdf/ciad313.pdf
- 2 Weeks of L-AmB: IV dose of 3 mg/kg of L-AmB for 2 weeks.
  https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10573726/pdf/ciad313.pdf
Arm/Group | Single Dose of L-AmB | 2 Doses of L-AmB | 2 Weeks of L-AmB
Number analyzed (Participants) | 38 | 36 | 38
Participants | 32 | 25 | 28

2. Secondary Outcome: Overall Mortality
Description: Mortality rates attributed to the cause of death that is not directly and only related to histoplasmosis
Time Frame: day 14
Population: Overall survival on day 14 were, respectively: 89.0% (34/38) (single-dose L-AmB-with 2 patients being excluded from efficacy analysis); 78.0% (29/37) (2-dose L-AmB arm-2 patients excluded from efficacy analysis); and 89.7% (35/38) (control group-1 patient excluded from efficacy analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of L-AmB | 2 Doses of L-AmB | 2 Weeks of L-AmB
Number analyzed (Participants) | 38 | 37 | 38
Participants | 4 | 8 | 3

ADVERSE EVENTS:
Time Frame: 14 days
Description: Kidney and liver toxicity - https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10573726/pdf/ciad313.pdf
Arm/Group | Single Dose of L-AmB | 2 Doses of L-AmB | 2 Weeks of L-AmB
All-Cause Mortality (participants affected / at risk) | 4/38 | 8/37 | 3/38
Serious Adverse Events (participants affected / at risk) | 1/38 | 6/37 | 4/38
Other Adverse Events (participants affected / at risk) | 34/38 | 27/37 | 34/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose of L-AmB (N=38) | 2 Doses of L-AmB (N=37) | 2 Weeks of L-AmB (N=38)
KDIGO (Renal and urinary disorders) | 1 (1) | 6 (6) | 4 (4) — Renal toxicity stage 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Single Dose of L-AmB (N=38) | 2 Doses of L-AmB (N=37) | 2 Weeks of L-AmB (N=38)
Infusion related toxicity (Blood and lymphatic system disorders) | 7/37 (7) | 5 (5) | 1 (1)
Hypokalemia (Renal and urinary disorders) | 3 (3) | 6 (6) | 12 (12) — Serum potassium levels of <3.5 mg/dL on day 14
Hemoglobin drop (Blood and lymphatic system disorders) | 7 (7) | 4 (4) | 8 (8) — Hemoglobin dropped >2 g/dL by day 14
Hypomagnesemia (Renal and urinary disorders) | 17 (17) | 12 (12) | 13 (13) — Serum magnesium levels of <1.8 mg/dL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT04059770/Prot_SAP_000.pdf